CLINICAL TRIAL: NCT01545765
Title: Anesthetic Effect Duration Produced by Lidocaine 7% + Tetracaine 7% Cream on 2 Different Body Areas
Brief Title: Anesthetic Effect Duration Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.03.SPR.29103
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2013-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lidocaine 7% and tetracaine 7% (Experimental)
  Interventions: Drug: Lidocaine 7% + Tetracaine 7% cream

INTERVENTIONS:
Drug: Lidocaine 7% + Tetracaine 7% cream — Study drug will be applied with a different application time to one side of the face and anterior thigh according to the randomization list.

SUMMARY:
The purpose of this study is to evaluate the duration of anesthetic effect produced , Lidocaine7% + Tetracaine 7% cream when applied with 2 different application times on the face and thigh.

DETAILED DESCRIPTION:
Subjects will have 4 target zones defined; 2 on the face and 2 on the anterior thighs. Upon inclusion into the study, subjects will have the study drug applied with a different application time to one side of the face and anterior thigh according to the randomization. After the completion of the application process, study drug on both sides of the face and on both anterior thighs will be removed by peeling.

After drug removal, the duration of anesthetic effect of the study drug will be tested using a pinprick test. Five (5) pinpricks using a 21-gauge needle will be performed at the 4 target zones (each side of the face and both anterior thighs). The pinprick test will be repeated up to 8 hours after drug removal. There will be a total of 20 post drug removal pinprick test completed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male of female subjects aged 18 or older with a normal not excessive hairy skin,

Exclusion Criteria:

* Female subjects who are pregnant or breast-feeding; or plan to become pregnant,
* Subjects who have a known allergy to one of the components of the test drug lidocaine, tetracaine or other local anesthetics,
* Subjects who are at risk in terms of precautions, warnings, and contra-indication with the study product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina YAVEL, MD- Dermatologist, Principal Investigator — Galderma investigational center
Locations (1):
- Galderma Investigational center, Rochelle Park, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 31 healthy volunteers have been enrolled in one Phase I center at USA.First subject in: May 3d 2012; Last subject ou: May 26th 2012.
Period: Overall Study
Arm/Group | Face 2 Application Times/ Thight 2 Application Times
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No sample size determination as a standard sample size for this type of study is about 30 subjects.
Arm/Group | Lidocaine 7% and Tetracaine 7%
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (1.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Secondary Outcome: Adverse Events
Description: Incidence of adverse events was to be reported during the study period
Time Frame: During the study
Population: A standard sample size for this type of study is 30 subjects. The analyses are performed on the safety population (APT), corresponding to the enrolled and randomized population, after exclusion of subjects who never applied the treatments with certainty. Missing data were to be treated as missing for all analyses.
Measure: Number; unit: participants
Arm/Group | Lidocaine 7% + Tetracaine 7% Face - First Application Time | Lidocaine 7% + Tetracaine 7% Face - Second Application Time | Lidocaine 7% + Tetracaine 7% Thigh - First Application Time | Lidocaine 7% + Tetracaine 7% Thigh - Second Application Time
Number analyzed (Participants) | 31 | 31 | 31 | 31
participants | 2 | 2 | 2 | 2

2. Primary Outcome: Duration of Anesthesia(Minutes)
Description: Onset and end of anesthesia are evaluated by Pinprick tests. Duration of anesthesia is calculated as: difference between onset and end of anesthesia (minutes).
Time Frame: From T0 (product removal) up to T8 hours after product removal
Population: as for outcome 1
Measure: Median (Full Range); unit: Minutes
Arm/Group | Lidocaine 7% + Tetracaine 7% Face - First Application Time | Lidocaine 7% + Tetracaine 7% Face - Second Application Time | Lidocaine 7% + Tetracaine 7% Thigh - First Application Time | Lidocaine 7% + Tetracaine 7% Thigh - Second Application Time
Number analyzed (Participants) | 31 | 31 | 31 | 31
Minutes | 80 [0 to 420] | 140 [0 to 480] | 0 [0 to 460] | 400 [0 to 480]

ADVERSE EVENTS:
Time Frame: All study period (from Baseline to end of teh study)
Description: Incidence of adverse events was to be reported during the study
Arm/Group | Lidocaine 7% + Tetracaine 7%
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine 7% + Tetracaine 7% (N=31)
SINUS HEADACHE (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitation or caveat on this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor to review and approval at least 2 months prior to the date of intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.